CLINICAL TRIAL: NCT00483067
Title: Phase II Study: 2-Chlorodeoxyadenosine (2-CdA) and Cytarabine (Ara-C) in Idiopathic Hypereosinophilic Syndrome (HES)
Brief Title: 2-Chlorodeoxyadenosine and Cytarabine in Patients With Idiopathic Hypereosinophilic Syndrome (HES)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-232
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: Idiopathic Hypereosinophilic Syndrome; Leukemia; 2-Chlorodeoxyadenosine; Cladribine; Cytarabine; Ara-C; 2-CdA; G-CSF; HES
MeSH Terms: conditions — Leukemia; Hypereosinophilic Syndrome | interventions — Cladribine; Cytarabine; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2-CdA + Ara-C + G-CSF (Experimental): 2-CdA 12 mg/m^2/day by vein (IV) Continuous Infusion and Ara-C 1 gm/m^2/day IV for 5 Days with G-CSF 5 mcg/kg/day subcutaneously starting Day 9
  Interventions: Drug: 2-CdA; Drug: Ara-C; Drug: G-CSF (Granulocyte colony-stimulating factor)

INTERVENTIONS:
Drug: 2-CdA — 12 mg/m^2/day by vein (IV) Continuous Infusion x 5 Days
  Other Names: 2-Chlorodeoxyadenosine; Cladribine
Drug: Ara-C — 1 gm/m^2/day IV Over 2 Hours x 5 Days
  Other Names: Cytarabine
Drug: G-CSF (Granulocyte colony-stimulating factor) — 5 mcg/kg/day given under the skin (subcutaneously) starting Day 9
  Other Names: Filgrastim; Neupogen; Granulocyte colony-stimulating factor; GCSF

SUMMARY:
Primary Objectives:

1. To determine the response rate, progression-free survival (PFS) and overall survival of patients who receive 2-CdA + Ara-C.
2. To examine if there is any clonality in the cytokine expression of helper T cells or cytokine receptor expression of eosinophils.
3. To determine the effect of 2-CdA on accumulation of Ara-C triphosphate in eosinophils.

DETAILED DESCRIPTION:
Before the study begins, patients will have a physical exam, blood tests, and urine tests. Women will have a pregnancy test. A bone marrow sample will be taken. This is done with a large needle. Heart tests and an MRI scan of the brain will be done if there is a suspicion of disease in the heart or central nervous system.

Patients in this study must have a catheter (thin tube) placed in a vein in the arm or under the collarbone. This tube will be left in place throughout the study. 2-CdA (Cladribine) will be given through the catheter 24 hours a day on days 2 to 6. Ara-C (Cytarabine) will be given through the catheter over 2 hours on days 1, 3, 4, 5, and 6. Starting on day 9, patients will inject G-CSF under their skin once a day; G-CSF helps blood counts return to normal. Treatment will be given on an inpatient or outpatient basis. The first course is normally done inpatient.

During the study, patients will have blood tests daily during the first week and every other day after that. Bone marrow samples will be taken on days 14, 21, and 28. Further bone marrow samples may be necessary to evaluate response. Heart tests and MRI scans of the brain may be done.

This is an investigational study. G-CSF, 2-CdA, and Cytarabine are approved by the FDA for treatment of cancer. Up to 40 patients will take part in this study. Patients will be treated at M. D. Anderson or other centers. A total of 40 people will take part in this study. About 1 patient every 3 months will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have diagnosis of idiopathic HES, defined as (1) no recent history of allergic reaction or parasitic infection; (2) sustained (> 6 months) hypereosinophilia (1,500/mm^3); and (3) signs or symptoms of organ involvement.
2. Age less than 76 years old.
3. Patient is not pregnant.
4. Zubrod performance status < 3.
5. Life expectancy is not severely limited by concomitant illness.
6. Serum creatinine < 2 mg/dL.
7. Serum bilirubin < 2 times upper limit of normal (2 mg/dL).
8. Alanine aminotransferase (SGPT) < 2 times upper limit of normal (112 IU/L).
9. Participant has completed the informed consent process, understands the investigational nature of the study, agrees to participate, and has signed the informed consent.

Exclusion Criteria:

1. Evidence of chronic active hepatitis or cirrhosis, and > 1 month from prior episode of hepatitis.
2. Presence of an active infection.
3. HIV positive.
4. Has eosinophilic leukemia (defined by presence of clonal cytogenetic abnormalities).
5. Recent history of parasite infection.
6. Recent history of allergic reaction.

Max Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1998-03; Primary Completion 2006-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Patient Outcomes at 6 Weeks | Baseline to 6 weeks timepoint (day 42)
  Patient outcomes defined at 6 weeks as Complete Remission (CR), absolute eosinophil count less than 1,500/mm3 and less than 5% of eosinophilic infiltrates in the bone marrow; and PR (partial response) defined as major clinical improvement without meeting the criteria specified for CR including an improvement in performance status to Zubrod's 0 or 1 along with clearance of clinical signs and symptoms of disease that are present at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Andreeff, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org